CLINICAL TRIAL: NCT00672022
Title: Pharmacokinetics, Safety and Tolerability of Zavesca (Miglustat) in Patients With Infantile Onset GM2 Gangliosidosis: Single and Steady State Oral Doses
Brief Title: Pharmacokinetics, Safety and Tolerability of Zavesca (Miglustat) in Patients With Infantile Onset Gangliosidosis: Single and Steady State Oral Doses
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Collaborators: Actelion (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3445
Record Dates: First submitted 2008-05-02; First posted 2008-05-06 (Estimated); Last update posted 2008-05-06 (Estimated); Status verified 2005-07

CONDITIONS: GM2 Gangliosidoses; Tay-Sachs; Sandhoff Disease
MeSH Terms: conditions — Gangliosidoses, GM2; Sandhoff Disease | interventions — miglustat

INTERVENTIONS:
Drug: Zavesca (Miglustat)

SUMMARY:
We want to see if Zavesca (or miglustat) is safe and can be tolerated by patients with acute infantile onset GM2 gangliosidosis - classical Tay-Sachs and infantile onset Sandhoff disease. We know that miglustat inhibits the formation of GM2 ganglioside, the compound that is stored in the brains of children with Tay-Sachs and Sandhoff disease. Since it inhibits the synthesis of ganglioside, miglustat may be able to reduce or delay the onset of clinical symptoms.

DETAILED DESCRIPTION:
Specific Aims

The primary objective of the study is to investigate the pharmacokinetics of ZAVESCA® (miglustat, OGT918), when given as a single dose and at steady state, in infantile patients with GM2 gangliosidosis. The secondary objectives are to evaluate the tolerability and safety of single and multiple doses of miglustat and to monitor disease progression using physical and developmental assessments and disease-specific biomarkers.

ELIGIBILITY:
Inclusion criteria

1. Diagnosis of GM2 gangliosidosis, confirmed by demonstration of profound deficiency of -hexosaminidase A or A & B in peripheral blood leukocytes or in cultured skin fibroblasts, within the previous 1 year in non-bone marrow transplant recipients who are < 2 years of age, or prior to stem cell transplant in stably engrafted transplant patients who are < 5 years of age.
2. Onset of characteristic clinical symptoms of the disease before the age of 9 months.
3. Normal renal and hepatic function.
4. Written informed consent from parent or legal guardian.

Exclusion criteria

1. Patients who are unable to comply with the study procedures of this protocol, including the refusal to swallow the food used to mask the taste of the study drug and whose parents are unwilling to administer the drug through a nasogastric or gastrostomy tube.
2. Patients receiving other investigational agents within 3 months of study initiation.
3. Patients who are anemic (hemoglobin < 11 g/dl, and/or hematocrit < 34%)
4. Patients who have a history of significant gastrointestinal disorders, including clinically significant diarrhea (>3 liquid stools per day for > 7 days), without definable cause within 3 months of baseline visit.
5. Patients with a high probability of dying during the 6-month assessment period of the study.
6. Patients who in the opinion of the investigator (for whatever reason) are thought to be unsuitable for the study.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2004-07; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Biomarkers (level of GM2 ganglioside, chitotriosidase activity, anti-GM2 antibodies) in plasma, serum and CSF will be measured at initial visit (run-in period), Week 13, and Week 25.

SECONDARY OUTCOMES:
Neurophysiologic Assessment - EEG and BEAR tests will be done at initial visit (run-in period), Week 13, and Week 25.
Ophthalmology Assessment - comparision of the "cherry-red" macula changes will be made at initial visit (run-in period) and Week 25.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia J TIfft, MD, PhD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States